CLINICAL TRIAL: NCT06533878
Title: (Part A) A Non-randomized, Open, Single-dose Escalation to Evaluate Tolerability and Safety of Single Oral Dose of HY209; (Part B) A Block-randomized, Double-blinded, Placebo-controlled, Multiple-dose Escalation to Evaluate Tolerability and Safety of Multiple Oral Doses of HY209 Phase 1 Clinical Trial in Healthy Volunteers
Brief Title: Evaluate Tolerability and Safety of HY209 in Healthy Volunteers
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Kukjeon Pharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: HY209-Tab01
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part A Dose Level 1 (Other): HY209 10 mg (1 tablet; 10 mg qd) fed, morning
  Interventions: Drug: HY-209
- Part A Dose Level 2 (Other): HY209 50 mg (1 tablet; 50 mg qd) fed, morning
  Interventions: Drug: HY-209
- Part A Dose Level 3 (Other): 1. HY209 100 mg (1 tablet; 100 mg qd) fed, morning
  2. HY209 100 mg (2 tablets; 50 mg bid) fed, morning, evening
  Interventions: Drug: HY-209
- Part A Dose Level 4 (Other): 1. HY209 200 mg (2 tablets; 200 mg qd) fasting, morning
  2. HY209 200 mg (2 tablets; 200 mg qd) fed, morning
  Interventions: Drug: HY-209
- Part A Dose Level 5 (Other): 1. HY209 300 mg (3 tablets; 300 mg qd) fasting, morning
  2. HY209 300 mg (3 tablets; 300 mg qd) fed, morning
  Interventions: Drug: HY-209
- Part A Dose Level 6 (Other): 1. HY209 400 mg (4 tablets; 400 mg qd) fasting, morning
  2. HY209 400 mg (4 tablets; 400 mg qd) fed, morning
  Interventions: Drug: HY-209
- Part B Dose Level 1 (Placebo Comparator): 1. HY209 150 mg (3 tablets; 50 mg tid) fed, morning, afternoon, evening
  2. HY209 placebo fed, morning, afternoon, evening
  Interventions: Drug: HY-209; Drug: HY-209 placebo
- Part B Dose Level 2 (Placebo Comparator): 1. HY209 200 mg (2 tablets; 200 mg qd) fed, morning
  2. HY209 placebo fed, morning
  Interventions: Drug: HY-209; Drug: HY-209 placebo
- Part B Dose Level 3 (Placebo Comparator): 1. HY209 200 mg (2 tablets; 100 mg bid) fed, morning, evening
  2. HY209 placebo fed, morning, evening
  Interventions: Drug: HY-209; Drug: HY-209 placebo
- Part B Dose Level 4 (Placebo Comparator): 1. HY209 300 mg (3 tablets; 100 mg tid) fed, morning, afternoon, evening
  2. HY209 placebo fed, morning, afternoon, evening
  Interventions: Drug: HY-209; Drug: HY-209 placebo

INTERVENTIONS:
Drug: HY-209 — Enteric coated tablet in the following colors: pink for 100 mg and yellow for 50 mg, and white for 10 mg
Drug: HY-209 placebo — Enteric coated tablet in the following colors: pink for 100 mg and yellow for 50 mg
  Arms: Part B Dose Level 1; Part B Dose Level 2; Part B Dose Level 3; Part B Dose Level 4

SUMMARY:
* Primary study objectives in Parts A and B To determine the Maximum Tolerable Dose(MTD) of the study drug (repeated or single dose).
* Endpoint: • Adverse event(AEs), including objective and subjective symptoms, after the IP dosing as well as physical examinations, vital signs, ECGs, and laboratory tests findings related to the IP dosing

  • Dose-limiting toxicities (DLTs)
* Justification for endpoints: The safety will be assessed comprehensively by performing safety assessment and evaluating relevant variables by dose group.

The tolerability will be assessed in DLT analysis set. In a first-in-human clinical trial, tolerability of the drug administered is usually assessed through determination of dose-limiting toxicity (DLT). An accurate dose proportionality of toxicity was not observed, but toxicity was found at high doses, not at low doses following IV and oral administrations, except transdermal treatment. Thus, a relationship between toxicity and doses was confirmed.

In addition, HY209 showed a dose dependence in some efficacy endpoints, including dose-dependent inhibition of release of Tumor Necrosis Factor(TNF)-α and Il-1β, key inflammation factors related to inflammatory bowel disease. Thus, evaluating the occurrence of DLTs through sequential dose escalation is determined appropriate to assess the tolerability and safety of HY209.

* Primary study objectives in Part A (Dose levels 4-6): To evaluate the effects of food on HY209 bioavailability (absorption rate and volume) following a single oral dose in healthy volunteers.
* Endpoint: PK of HY209 at a fasting condition and after a high-fat meal Point estimates for the geometric mean ratio of variables (Area under concentration-time curve;AUC₀-₆, AUCₗₐₛₜ, AUC₀-∞, and Cmax) and the 90% confidence interval(CI) and Tmax .
* Justification for endpoints: For oral drugs, effects of food on bioavailability of the drugs are usually evaluated. Especially, a systemic exposure to bile acid drugs of enterohepatic circulation can be explained with a spillover from the liver to systemic circulatory system. Thus, a systemic exposure is thought to be affected by food, but the actual effects of food are triggered by combination of factors that affect in vivo elution of a drug and absorption of the active pharmaceutical ingredient(API) of the drug. As estimating the extent of effects on bioavailability is difficult without conducting an actual food effect study, there is a need for clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have received a full explanation about the study and the characteristics of the investigational product (IP), understood them, and then have provided voluntary consent for the study participation and fulfillment of the subject obligations during the study
2. Healthy adult males ≥ 19 years and ≤ 45 years of age at the time of screening
3. Subjects with weight ≥ 55 kg and ≤ 90 kg and BMI ≥ 18.0 and < 30.0 kg/m²
4. Subjects without congenital or chronic diseases and pathological symptoms or findings in the medical examinations
5. Subjects determined eligible for the study participation based on the results from laboratory tests, including serology, hematology, blood chemistry, urinalysis, and urine drug screening, vital signs, physical examinations, and electrocardiography (ECG), performed depending on the drug characteristics at screening (subjects with physical examinations, laboratory tests and ECG findings beyond the normal range may be allowed to take part in the study when they do not have clinically significant diseases and obvious ground for participation can be provided in the investigator's opinion)

Exclusion Criteria:

1. Clinically significant diseases or past history that precludes the study participation in the investigator's opinion
2. Occurrence of any diseases (illnesses) within 1 week prior to start of the IP dosing [e.g., flu epidemic or common cold, fever ≥ 38℃]). (However, when the disease is resolved in a short period of time, their study participation can be determined through a follow-up test after treatment.)
3. Unable or unwilling to take tablets
4. The following diseases and health conditions that may affect the pharmacokinetics (PK) of the IP, including absorption

   1. Gastrointestinal (GI) diseases (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.)
   2. Past history of cholecystectomy, bariatric procedures and/or any GI surgery that may interfere with the PK profile of the study drug, except simple cholecystectomy or hernia surgery
5. Rare hereditary problems of galactose intolerance, the Lapp lactose deficiency, or glucose galactose malabsorption
6. The following laboratory test results at screening (However, for liver tests, any test results that are considered to be caused by clinically meaningless transient changes or one-time alcohol consumption and night-shift work and other lifestyle can be finally confirmed through follow-up tests after the correction)

   1. Elevated alanine aminotransferase (ALT) > 1.1 x upper limit of normal (ULN)
   2. Elevated aspartate aminotransferase (AST) > 1.2 x ULN
   3. Elevated total bilirubin > 1.2 x ULN
   4. Elevated creatinine > 0.1 mg/dL from the ULN
   5. Estimated glomerular filtration rate(eGFR) < 60 mL/min/1.73 m²
7. Systolic blood pressure (BP) ≥ 150 mmHg or ≤ 100 mmHg, or diastolic BP ≥ 100 mmHg or ≤ 60 mmHg in the vital signs as measured in a sitting position after taking a rest for at least 3 minutes
8. Pulse rate < 50 beats/min (bpm) or > 90 bpm when measured in a sitting position after taking a rest for at least 3 minutes; or < 45 bpm when (1) a normal thyroid function is confirmed with interview, physical examinations, and Thyroid stimulating Hormone(TSH) tests and (2) there is no clinical symptom of bradycardia (orthostatic hypotension and vertigo).
9. Patients with clinically significant arrhythmia in the ECGs in the investigator's opinion (not applicable for the first degree atrioventricular(AV) block associated with the heart rate that meet the inclusion criteria)
10. Clinically significant findings in 12-lead ECGs at screening
11. History of malignancy, except for the following cases

    1. At least 5 years have passed without recurrence after appropriate treatments
    2. Appropriately treated thyroid cancer (papillary, follicular, and medullary types of Stage I or II), skin basal cell or squamous cell carcinoma and lentigo maligna (malignant black spots), and intraepithelial carcinoma in other areas
12. Patients with the following active infections:

    1. Tuberculosis (when confirmed with medical history, physical examinations, or radiological findings if needed, or Tuberculin(TB) test)
    2. Hepatitis B (perform hepatitis B surface(HBs) Ag only as screening; when confirmed positive in immunoglobulin M(IgM) anti-hepatitis B core antigen(HBc) and Hepatitis B virus(HBV) Nuclei acid test(NAT) tests)
    3. Hepatitis C (perform Anti-HCV only as screening; subjects with positive anti-HCV can take part in the study when negative result is confirmed in NAT for HCV RNA)
    4. HIV infection (Anti-HIV only for screening)
    5. Syphilis (perform venereal disease research laboratory(VDRL) or Rapid plasma reagin(RPR) as screening; patients with positive serology are not eligible)
13. Persistent alcohol consumption within 6 months prior to the first dose (exceeding 21 units/week, 1 unit = 10 g = 12.5 mL of pure alcohol) or unable to abstain from consuming alcohol throughout the study period from 72 hours prior to the first dose of the study drug to the end of study (the final visit) [e.g., 1 cup (250 mL) of beer (5%) = 1 glass (50 mL) of 10 g soju (20%) = 1 glass (125 mL) of 8 g wine (12%) = 12 g]
14. Smokers (subjects who quit smoking at least 6 months prior to screening and have negative urine cotinine test at screening or who have never smoked are eligible)
15. Whole blood donation or loss of substantial amount of blood within 2 months or apheresis within 1 month, or blood transfusion within 1 month prior to the first dose
16. Past history of hypersensitivity to any components of the IP
17. Subjects who have received any of the following drugs prior to the study participation and the required washout period has not passed

    1. Prescription or over-the-counter drugs: Periodic treatment with any prescription or over-the-counter drugs (including Vitamins). Subjects should discontinue the drugs at least 14 days prior to the first dose of the study drug. Subjects who want to take part in the study should discontinue any prescribed drugs upon the physician's decision.
    2. Oriental medications, herbal products, and dietary supplements: Subjects should discontinue use of herbal products or dietary supplements [e.g., St. John's Wort, ginseng, ginkgo biloba, and garlic supplements)] at least 14 days prior to the first dose of the study drug.
    3. Special fruits: Intake of grapefruit or grapefruit juice, Seville oranges, or pomelos should be restricted from at least 14 days prior to the first dose of the study drug.
18. History of substance or alcohol abuse or addiction within 2 years prior to the start of the study drug or positive screening results for alcohol, smoking, or abusive drugs [e.g., cotinine, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine or opioids, tricyclic antidepressants] at screening
19. Males who do not agree to use effective contraceptions during the study period and up to 3 months after the last dose of the study drug
20. Persons who do not agree to refrain from donating their sperms during the study period and at least 3 months after the last dose of the study drug
21. Persons who answer "Yes" to any of the questions in the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past 12 months at screening (for Part B only)
22. Persons who are participating in another clinical study or have taken a drug in another clinical study or bioequivalence study within 6 months prior to the first dose of the study drug (however, to determine the end of other study participation, the next day of the last dose will be counted as Day 1.)
23. Other cases that make the subject ineligible for the study

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 59 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events, physical examinations, vital signs, ECGs, laboratory tests findings related to the IP dosing, Does limiting toxicity, PK assessment endpoints | Test of DLTs observed until 7 days after the last does of HY209 for each dose and dosage cohort.
  Part A
  * AEs, including objective and subjective symptoms, after the IP dosing as well as physical examinations, vital signs, ECGs, and laboratory tests findings related to the IP dosing
  * [Part A: Phase 1a or Phase 1 dose escalation] incidence and frequency of DLTs observed until 7 days after HY209 treatment for each dose and dosage cohort
  * [Part A (Dose levels 4-6): effects of food on bioavailability] point estimates of geometric mean ratio for PK parameters (AUC₀-₆, AUCₗₐₛₜ, AUC₀-∞, and Cmax) following a single dose at a fasting condition and after a high-fat meal and the 90% CI and Tmax
  Part B
  * AEs, including objective and subjective symptoms, after the IP dosing as well as physical examinations, vital signs, ECGs, and laboratory tests findings related to the IP dosing
  * [Part B: Phase 1b or Phase 1 cohort expansion] incidence and frequency of DLTs observed until 7 days after the last dose of HY209 for each dose and dosage cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Kukjeon Pharmaceutical Co., Ltd., Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Zhong M. TGR5 as a Therapeutic Target for Treating Obesity. Curr Top Med Chem [Internet] 2010 [cited 2021 May 10];10(4):386-96. — http://pubmed.ncbi.nlm.nih.gov/20180762/
- See also: Chang S, Kim YH, Kim YJ, Kim YW, Moon S, Lee YY, et al. Taurodeoxycholate increases the number of myeloid-derived suppressor cells that ameliorate sepsis in mice. Front Immunol [Internet] 2018 [cited 2021 May 20];9(SEP):1984. — http://www.frontiersin.org
- See also: Kim H, Fang S. Crosstalk between FXR and TGR5 controls glucagon-like peptide 1 secretion to maintain glycemic homeostasis. Lab Anim Res [Internet] 2018 [cited 2021 May 26];34(4):140. — https://pubmed.ncbi.nlm.nih.gov/30671099/
- See also: Altman DG, Bland JM. Statistics notes. Treatment allocation in controlled trials: why randomise? BMJ [Internet] 1999 [cited 2016 Aug 30];318(7192):1209. — http://www.ncbi.nlm.nih.gov/pubmed/10221955
- See also: Pai D, Woo J-M, Son MH, Lee C. The Reliability and Validity of the Korean Version of ColumbiaSuicide Severity Rating Scale in Alcohol Dependent Patients. J Korean Neuropsychiatr Assoc [Internet] 2015 [cited 2019 Jun 21];54(2):222-7. — http://dx.doi.org/10.4306/jknpa.2015.54.2.222
- See also: Svedlund J, Sjödin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci [Internet] 1988 [cited 2017 Jul 18];33(2):129-34. — http://www.ncbi.nlm.nih.gov/pubmed/3123181
- See also: Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res [Internet] 1998 [cited 2017 Jul 18];7(1):75-83. — http://www.ncbi.nlm.nih.gov/pubmed/9481153
- See also: Monés J, Adan A, Segú JL, López JS, Artés M, Guerrero T. Quality of life in functional dyspepsia. Dig Dis Sci [Internet] 2002 [cited 2017 Jul 18];47(1):20-6. — http://www.ncbi.nlm.nih.gov/pubmed/11837724
- See also: Wiklund IK, Fullerton S, Hawkey CJ, Jones RH, Longstreth GF, Mayer EA, et al. An irritable bowel syndrome-specific symptom questionnaire: development and validation. Scand J Gastroenterol [Internet] 2003 [cited 2017 Jul 18];38(9):947-54. — http://www.ncbi.nlm.nih.gov/pubmed/14531531